CLINICAL TRIAL: NCT03009136
Title: Efficacy and Safety of So-Cheong-Ryong-Tang on Perennial Allergic Rhinitis: Study Protocol for a Double-blind, Randomized, Parallel-group, Multi-center Trial
Brief Title: Efficacy and Safety of So-Cheong-Ryong-Tang on Perennial Allergic Rhinitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Collaborators: Kyung Hee University Hospital (Other); Pusan National University Hospital (Other); Semyung University Affiliated Oriental Medical Hospital (Other); DongGuk University (Other)
Responsible Party: Principal Investigator, Minhee Kim, Clinical Professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISEE_2015_SCRT
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Perennial Allergic Rhinitis; Herbal Medicine; Korean Medicine; So-Cheong-Ryong-Tang
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCRT group (Experimental): 3g, three times a day, each taken before or between meals
  Interventions: Drug: SCRT
- placebo group (Placebo Comparator): 3g, three times a day, each taken before or between meals
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: SCRT — composed of eight herbs: Glycyrrhiza uralensis Fischer 1g Zingiber officinale Roscoe 0.5g Cinnamomum cassia Blume 0.2g, Ephedra sinica Stapf 0.5g, Pinellia ternata Breitenbach 2.67g, Paeonia lactiflora PALL 1g, Asiasarum sieboldi F. Maekawa 0.5g, Schisandra chinensis 2.67g (per 9g of granules)
  Arms: SCRT group
Drug: Placebos — is made of lactose, corn starch and caramel coloring, and has appearance, shape, weight, taste, and color similar to SCRT
  Arms: placebo group

SUMMARY:
The aim of this study is to investigate the short and long term efficacy and the safety of SCRT treatment for PAR

ELIGIBILITY:
Inclusion Criteria:

1. age 18-60 years
2. presence of two or more nasal symptoms (rhinorrhea, nasal congestion, nasal itching and sneezing) with severity score ≥ 2 (0 = no symptom, 1 = mild symptom, 2 = moderate symptom, and 3=severe symptom)
3. presence of nasal symptoms more than 2 consecutive years; and
4. positive reaction to the one or more perennial allergen in skin prick test.

Exclusion Criteria:

1. treatment with nasal/oral corticosteroids within the past month; nasal cromolyn or tricyclic antidepressants within the past two weeks; or nasal/oral decongestants, nasal/oral antihistamines, or antileukotrienes within the past week
2. presence of rhinosinusitis (paranasal sinus X-ray demonstrating mucosal thickening, or partial or complete opacification of the paranasal sinuses)
3. presence of hypertension (systolic ≥ 180 mmHg or diastolic ≥ 100 mmHg)
4. presence of abnormal liver function (aspartate transaminase (AST) or alanine transaminase (ALT) ≥ 100 IU/L) or abnormal renal function (blood urea nitrogen (BUN) ≥ 30 mg/dL or creatinine ≥ 1.8 mg/dL (male), 1.5 mg/dL (female))
5. presence of neoplasm, severe systemic inflammation, other systemic disease that affects rhinitis
6. history of drug allergy
7. history of anaphylaxis for allergic tests
8. pregnancy or lactation
9. participation of other clinical study within the past 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2016-12-31 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Total Nasal Symptom score | At baseline, week 2, 4, 8, 12

SECONDARY OUTCOMES:
Change from baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) score | At baseline, week 2, 4, 8, 12
Change from baseline in Total serum IgE level | At baseline, week 4
Change from baseline in eosinophil count | At baseline, week 4
Change from baseline in cytokine level | At baseline, week 4

CONTACTS AND LOCATIONS:
Overall Officials: Minhee Kim, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim MH, Ko Y, Ahn JH, Yun Y, Yun MN, Ko SG, Choi I. Efficacy and safety of So-Cheong-Ryong-Tang in treatment of perennial allergic rhinitis: study protocol for a double-blind, randomised, parallel-group, multicentre trial. BMJ Open. 2017 Sep 27;7(9):e016556. doi: 10.1136/bmjopen-2017-016556. PMID 28963290